CLINICAL TRIAL: NCT04029168
Title: Pelvic Floor Muscles Efficiency as an Independent Factor of Therapeutic Success in the Surgical Treatment of Stress Urinary Incontinence and Pelvic Organ Prolapse
Brief Title: Pelvic Floor Muscles and Success in the Surgical Treatment of Stress Urinary Incontinence and Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PN/25/2019
Record Dates: First submitted 2019-07-09; First posted 2019-07-23 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Stress Urinary Incontinence; Pelvic Organ Prolapse; Pelvic Floor Disorders
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Organ Prolapse; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pelvic floor surgery: The group will consist of females with pelvic floor disorders (pelvic organ prolapse, stress urinary incontinence) qualified for pelvic floor surgery

SUMMARY:
The aim of the study is evaluation of the efficiency of pelvic floor muscles in the context of surgical outcomes in the treatment of stress urinary incontinence and pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal and postmenopausal women
* stress urinary incontinence
* pelvic organ prolapse

Exclusion Criteria:

- previous surgical interventions due to stress urinary incontinence or pelvic organ prolapse

Ages: 30 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Study Population: Women with stress urinary incontinence and pelvic organ prolapse
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory (PFDI-20) | change from the baseline till 6 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic floor organ prolapse quantification (POP-Q) | change from the baseline till 6 month post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Marshall-Bonney test | change from the baseline till 6 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory (PFDI-20) | 3 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic Floor Distress Inventory (PFDI-20) | 12 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic Floor Distress Inventory (PFDI-20) | change from the baseline till 3 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic Floor Distress Inventory (PFDI-20) | change from the baseline till 12 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Visual Analogue Scale | 3 month post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
Visual Analogue Scale | 6 months post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
Visual Analogue Scale | 12 months post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
Visual Analogue Scale | change from the baseline till 3 months post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
Visual Analogue Scale | change from the baseline till 6 months post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
Visual Analogue Scale | change from the baseline till 12 months post treatment
  Distress assessment range 0-10, higher numbers represent better outcomes
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | 3 month post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | 6 months post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | 12 months post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | change from the baseline till 3 months post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | change from the baseline till 6 months post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
PELVIC FLOOR IMPACT QUESTIONNAIRE SHORT FORM (PFIQ-7) | change from the baseline till 12 months post treatment
  Assessment of life impact in women with pelvic floor disorders, range 0-300, higher numbers indicate greater impact
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | 3 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | 6 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | 12 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | change from the baseline till 3 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | change from the baseline till 6 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Incontinence impact Questionnaire-Short Form (IIQ-7 SF) | change from the baseline till 12 months post treatment
  To measure the impact of urinary incontinence on activities, roles and emotional states
Pelvic floor organ prolapse quantification (POP-Q) | at 1 month post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Pelvic floor organ prolapse quantification (POP-Q) | 3 months post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Pelvic floor organ prolapse quantification (POP-Q) | 12 months post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Pelvic floor organ prolapse quantification (POP-Q) | change from the baseline till 3 month post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Pelvic floor organ prolapse quantification (POP-Q) | change from the baseline till 12 month post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Pelvic floor organ prolapse quantification (POP-Q) | change from the baseline till 1 month post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Marshall-Bonney test | at 1 month post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Marshall-Bonney test | 3 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Marshall-Bonney test | 12 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Marshall-Bonney test | change from the baseline till 3 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Marshall-Bonney test | change from the baseline till 1 month post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Marshall-Bonney test | change from the baseline till 12 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence
Pelvic Floor Distress Inventory (PFDI-20) | 6 months post treatment
  Symptom inventory and a measure of the degree of bother and distress. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic floor organ prolapse quantification (POP-Q) | 6 months post treatment
  Quantification of pelvic organ prolapse, range 0-4, higher indicate worse outcomes
Marshall-Bonney test | 6 months post treatment
  Assessment of stress urinary incontinence, test can be negative or positive, positive test indicates incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Sys, PhD, Study Chair — Centre of Postgraduate Medical Education
Locations (1):
- Centrum Medyczne "ŻELAZNA", Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided